CLINICAL TRIAL: NCT03638531
Title: Long-Term Transcranial Direct Current Stimulation in Parkinson's Disease
Brief Title: Long- Term Transcranial Direct Current Stimulation in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Brach Poston, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002548
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
Keywords: tDCS; cortical excitability; motor cortex; motor learning; handwriting; micrographia
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): Anodal tDCS will be applied in nine experimental sessions over a 2-week period.
  Interventions: Device: Anodal tDCS
- SHAM tDCS (Sham Comparator): SHAM tDCS will be applied in nine experimental sessions over a 2-week period.
  Interventions: Device: SHAM tDCS

INTERVENTIONS:
Device: Anodal tDCS — Anodal tDCS will be applied over the FDI muscle representational area of the motor cortex for 25 minutes in combination with the two motor tasks (precision grip task and handwriting task).
  Arms: Anodal tDCS
Device: SHAM tDCS — SHAM tDCS will be applied over the FDI muscle representational area of the motor cortex for 25 minutes in combination with the two motor tasks (precision grip task and handwriting task).
  Arms: SHAM tDCS

SUMMARY:
The goal of the proposed research is to determine the influence of transcranial direct current stimulation (tDCS) on long-term motor learning, transfer of motor learning, and cortical function in Parkinson's disease (PD). The project comprises a 2 week training study that will involve tDCS applied during two practice motor tasks with behavioral, clinical, and physiological evaluations at baseline as well as 1, 14 and 28 days following the 2 week training and stimulation period. The findings of the proposed studies should have significant clinical significance and applications to comprehensive intervention therapy development in the treatment of PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and affects approximately 1 million people in the United States with total annual costs approaching 11 billion dollars. Current medical and surgical treatment approaches for PD are either only mildly effective, expensive, or associated with a variety of side effects. Therefore, the development of practical and effective therapeutic adjuncts to current treatment approaches would have significant benefits.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate cortical excitability and improve motor function in healthy subjects, older adults, and in stroke. However, there are several crucial issues that currently prevents the determination of the viability of tDCS as an adjunct intervention in PD. For example, the magnitude to which tDCS may be able to improve long-term motor learning beyond what can be achieved by practice alone in PD is unknown. It is also unclear if short-term improvements in motor function induced by tDCS and measured in the OFF state in PD can be attained over the long-term in the ON state, which is necessary for real world application. In addition, it is uncertain if the effects of tDCS generalize to non-practiced tasks and to the ipsilateral, non-tDCS stimulated hand. Finally, the physiological mechanisms underlying any of these issues have not been identified because no long-term motor learning tDCS studies in PD to date have concurrently quantified behavioral, clinical, and physiological measures.

The project will be a single-center, double-blind, randomized, sham-controlled, experimental design. PD patients will practice 2 motor tasks (practice tasks) with their right (primarily affected) hand in 9 practice sessions over a 2 week period in association with either tDCS or SHAM stimulation of the left (contralateral) motor cortex. In addition, 4 testing sessions will be performed and will include a Baseline test, an end of training test (EOT), a follow up test 2 weeks after the end of training (EOT+14), and a follow up test 4 weeks after the end of training (EOT+28). The primary outcome variables will be the force error in the first practice task (precision grip task; PGT) and the stroke amplitude, stroke variability, and writing speed in the second practice task (handwriting task; HWT). The secondary outcome variables the Unified Parkinson's Disease Rating Scale (UPDRS) Part 3, the Purdue Pegboard Test (PT), and the Jebsen Taylor Hand Function Test (JTT).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent.
2. A clinical diagnosis of idiopathic PD.
3. A stable and optimal medical regimen of anti-parkinsonian drug therapy for the duration of the study.
4. Modified Hoehn and Yahr stage between 1.0 and 3.0 in the OFF state.
5. Right-hand dominant and primarily right-side affected to prevent confounds due to handedness and affected side.

Exclusion Criteria:

1. An uncontrolled medical condition (i.e. hypertension, diabetes, etc).
2. Evidence of secondary or atypical parkinsonism as suggested by:

   1. History of CVA's, exposure to toxins, neuroleptics or encephalitis.
   2. Neurologic signs of upper motor neuron or cerebellar involvement, supranuclear gaze palsy or significant orthostatic hypertension.
3. Metal in the skull or the eye, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, and metal fragments in the eye, as these may make TMS and tDCS unsafe.
4. An uncertainty about the presence of metal objects in a subject's body exists.
5. Hearing loss, have had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures, have another neurological disorder other than a movement disorder, or have a head injury where they passed out for more than a few seconds.
6. Pregnant or thought to be pregnant.
7. Irrepressible dyskinesia or tremor to prevent the confound of excessive EMG during TMS testing at rest.
8. Any other neurological disorders.
9. Meeting of any of the TMS exclusion criteria given in international guidelines.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Force error in the precision grip task | Baseline, 1 day post, 2 weeks post, 4 weeks post
  Changes in force error after the two week intervention
Handwriting task performance | Baseline, 1 day post, 2 weeks post, 4 weeks post
  Changes in stroke amplitude, stroke variability, and writing speed after the two week intervention

SECONDARY OUTCOMES:
Transfer of motor learning | Baseline, 1 day post, 2 weeks post, 4 weeks post
  Changes in the UPDRS Motor Section Part 3 after the two week intervention
Transfer of motor learning | Baseline, 1 day post, 2 weeks post, 4 weeks post
  Changes in the Purdue Pegboard Test after the two week intervention
Transfer of motor learning | Baseline, 1 day post, 2 weeks post, 4 weeks post
  Changes in the Jebsen Taylor Hand Function Test after the two week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brach Poston, Ph.D., Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- Bigelow Health Sciences, Las Vegas, Nevada, United States